CLINICAL TRIAL: NCT04759924
Title: Skin Structure, Skin Function and Skin Microbiome of Pregnant Females and Their Newborns: a Descriptive Longitudinal Study
Brief Title: Mother - Newborn Observational Study
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ulrike Blume-Peytavi, MD, Head of Clinical Research Center for Hair and Skin Science, Charite University, Berlin, Germany
Other Study IDs: CRC-SP-AC-38
Record Dates: First submitted 2021-02-03; First posted 2021-02-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Skin Microbiome
Keywords: descriptive longitudinal study; skin structure; skin function; skin microbiome; hair growth; pregnancy; newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab of the skin microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pregnancy leads to a number of skin changes but empirical evidence about the structural and functional changes of the skin is scarce. Findings on skin structure and function in newborns and children in the first year of life reveal a rapid skin maturation after birth, but evidence indicates, that in particular water-holding and transport mechanisms are very different to adults in the first year in life. The most important open question is whether and how the maternal cutaneous properties predict the skin function of their children. This is especially relevant for the skin microbiome, because it closely interacts with the host and is assumed to play a role in many skin diseases. Therefore, the objective of this study is the description of characteristics of skin and hair structure and skin function of pregnant women and their newborns during pregnancy and for both in the first six months after delivery. In addition, we investigate associations of the mother's and their newborns skin microbiomes, and changes thereof in the newborns within the first six months of life.

The study has a descriptive, exploratory, longitudinal design. We will recruit pregnant females between 18 to 45 years old using advertisement campaigns, study information material in the waiting areas of their gynecologists, in pregnancy preparation services and in hospital's outpatient services. If they are interested and fulfill the inclusion criteria, they are invited to participate. Taking into account an assumed dropout rate of about 30%, a final sample of n = 100 women is expected. A detailed dermatological examination and general medical condition are documented. Non-invasive, standardized skin and hair physiological and skin microbiome measurements are performed during the visits. Baseline is scheduled during pregnancy until late 4 weeks before delivery. Follow-up visits are scheduled 4 weeks and 6 months after birth for mothers and newborns. Descriptive statistical methods will be calculated for frequencies and associations over time depending on scale levels of the measurements.

In our longitudinal study, we will characterize a broad range of individual and environmental characteristics of mothers and their newborns to evaluate interrelationships with skin parameters and their changes over the period of at least 8 months. Considering these multiple variables and levels together will allow a deeper understanding of the complex interrelationship of the newborns skin maturation.

DETAILED DESCRIPTION:
A longitudinal descriptive, exploratory cohort study will be performed including females during pregnancy, puerperium and their newborns until sixth months of life.

Women will be invited after the first pregnancy trimester from the federal state of Berlin (Germany) during their visits to gynecologists and/or midwives. Inclusion and all study visits and measurement procedures will be conducted at the Clinical Research Center for Hair and Skin Science at the Department of Dermatology at the Charité-Universitätsmedizin Berlin (Germany). If meeting the eligibility criteria women will be included into the study. After inclusion into the study during the baseline visit, women will be followed at date of delivery + four weeks and followed further at the sixth month after delivery. The newborn/infants will be examined up to four weeks after birth and will be followed at sixth month after birth.

Due to the descriptive and exploratory nature of this study a broad range of characteristics and variables will be measured. Main aspects are skin structure, skin function and skin microbiome in one skin area. Skin structure will be measured by means of skin surface topography, epidermal thickness, skin stiffness and elasticity. Skin function will be measured by means of stratum corneum hydratation (SCH), TEWL and skin surface pH, which are established parameters to characterize the skin barrier function. Skin microbiome is defined as bacterial diversity, in detail the relative abundance of phylotypes, operational taxonomic units (OTU) will be measured. Hair growth will be measured on central and occipital scalp by means of hair density, hair widths.

ELIGIBILITY:
Inclusion criteria

* written informed consent
* clinically healthy skin and hair appearance
* being free of any dermatological condition
* acceptance to abstain from sunbathing
* acceptance to abstain from solarium
* agreement to use the same skin cleaning and caring procedures during the study

Exclusion Criteria:

* regular smoking
* regular alcohol intake
* any dermatological condition or skin affection which may interfere with the study assessments (psoriasis, atopic dermatitis or other lesions at the investigational sites)
* clinically significant, possibly unstable medical conditions due to gravidity such as gestosis, eclampsia or thrombosis.
* Criteria related to treatments and products such as current topical or systemic treatment possibly affecting the skin, (diuretics, cholesterol-lowering drugs, hormones) during past four weeks
* therapeutic ultraviolet radiation within six weeks before inclusion
* increased ultraviolet-exposure within six weeks before inclusion

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women and their newborns
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline stratum corneum hydratation (SCH) at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  measurement of skin hydration: arbitrary units 0-120 , whereas higher readings indicate higher stratum corneum hydration
Change from baseline Skin surface pH at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  Skin pH-meter measurement (range from 4 to 7,5)
Change from baseline Transepidermal water loss (TEWL ) at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  Transepidermal waterloss through the stratum corneum in g per hour per m2 (range: 0,0-60,0 g/m2/h)
Change from baseline Skin stiffness and elasticity at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  total extensibility (Uf, mm), Structural elasticity Uf) of the skin (0,00-0,50 Uf in mm/degree)
Change from baseline Epidermal thickness at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  Standardized images via Optical coherence tomography (OCT) measured in mm
Change from baseline Skin surface topography at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  Standardized images via Visioscan
  * RA (arithmetic mean roughness) in µm
  * RZ (arithmetic mean roughness from five sampling length) in µm
Change from baseline Skin microbiome at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  Bacterial diversity Relative abundance of phylotypes (operational taxonomic units, (OTUs)
Change from baseline Hair growth at 4 weeks and 6 months after delivery | baseline visit mother at least 4 weeks before delivery, mother and newborn: 4 weeks and 6 months after delivery
  Measurement of Hair thickness

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Prof. MD, Principal Investigator — Charité Universitätsmedizin Berlin, Klinik für Dermatologie, Venerologie und Allergologie
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Surber C, Dragicevic N, Kottner J. Skin Care Products for Healthy and Diseased Skin. Curr Probl Dermatol. 2018;54:183-200. doi: 10.1159/000489532. Epub 2018 Aug 21. PMID 30130786
- [Background] Muallem MM, Rubeiz NG. Physiological and biological skin changes in pregnancy. Clin Dermatol. 2006 Mar-Apr;24(2):80-3. doi: 10.1016/j.clindermatol.2005.10.002. PMID 16487877
- [Background] Vora RV, Gupta R, Mehta MJ, Chaudhari AH, Pilani AP, Patel N. Pregnancy and skin. J Family Med Prim Care. 2014 Oct-Dec;3(4):318-24. doi: 10.4103/2249-4863.148099. PMID 25657937
- [Background] Panicker VV, Riyaz N, Balachandran PK. A clinical study of cutaneous changes in pregnancy. J Epidemiol Glob Health. 2017 Mar;7(1):63-70. doi: 10.1016/j.jegh.2016.10.002. Epub 2016 Nov 19. PMID 27870929
- [Background] Ciechanowicz P, Sikora M, Taradaj K, Ruta A, Rakowska A, Kociszewska-Najman B, Wielgos M, Rudnicka L. Skin changes during pregnancy. Is that an important issue for pregnant women? Ginekol Pol. 2018;89(8):449-52. doi: 10.5603/GP.a2018.0077. PMID 30215465
- [Background] Martins-Costa GM, Bakos R. Total Body Photography and Sequential Digital Dermoscopy in Pregnant Women. Dermatol Pract Concept. 2019 Apr 30;9(2):126-131. doi: 10.5826/dpc.0902a08. eCollection 2019 Apr. PMID 31106015
- [Background] Thom E. Pregnancy and the hair growth cycle: anagen induction against hair growth disruption using Nourkrin(R) with Marilex(R) , a proteoglycan replacement therapy. J Cosmet Dermatol. 2017 Sep;16(3):421-427. doi: 10.1111/jocd.12286. Epub 2016 Sep 23. PMID 27659896
- [Background] Pierard-Franchimont C, Pierard GE. Alterations in hair follicle dynamics in women. Biomed Res Int. 2013;2013:957432. doi: 10.1155/2013/957432. Epub 2013 Dec 24. PMID 24455742
- [Background] Boyer G, Lachmann N, Bellemere G, De Belilovsky C, Baudouin C. Effects of pregnancy on skin properties: A biomechanical approach. Skin Res Technol. 2018 Nov;24(4):551-556. doi: 10.1111/srt.12465. Epub 2018 Feb 26. PMID 29479745
- [Background] Ludriksone L, Garcia Bartels N, Kanti V, Blume-Peytavi U, Kottner J. Skin barrier function in infancy: a systematic review. Arch Dermatol Res. 2014 Sep;306(7):591-9. doi: 10.1007/s00403-014-1458-6. Epub 2014 Mar 5. PMID 24595645
- [Background] Nikolovski J, Stamatas GN, Kollias N, Wiegand BC. Barrier function and water-holding and transport properties of infant stratum corneum are different from adult and continue to develop through the first year of life. J Invest Dermatol. 2008 Jul;128(7):1728-36. doi: 10.1038/sj.jid.5701239. Epub 2008 Jan 17. PMID 18200056
- [Background] Visscher MO, Adam R, Brink S, Odio M. Newborn infant skin: physiology, development, and care. Clin Dermatol. 2015 May-Jun;33(3):271-80. doi: 10.1016/j.clindermatol.2014.12.003. Epub 2014 Dec 8. PMID 25889127
- [Background] Oranges T, Dini V, Romanelli M. Skin Physiology of the Neonate and Infant: Clinical Implications. Adv Wound Care (New Rochelle). 2015 Oct 1;4(10):587-595. doi: 10.1089/wound.2015.0642. PMID 26487977
- [Background] Hughes-Formella B, Wunderlich O, Williams R, Fernandez J, Kim YZ, Wigger-Alberti W, Pecquet S, Moodycliffe A. Comparison of Skin Structural and Functional Parameters in Well-Nourished and Moderately Undernourished Infants. Skin Pharmacol Physiol. 2019;32(4):212-223. doi: 10.1159/000499434. Epub 2019 Jun 5. PMID 31167217
- [Background] Fluhr JW, Darlenski R. Skin Surface pH in Newborns: Origin and Consequences. Curr Probl Dermatol. 2018;54:26-32. doi: 10.1159/000489515. Epub 2018 Aug 21. PMID 30130770
- [Background] Findley K, Grice EA. The skin microbiome: a focus on pathogens and their association with skin disease. PLoS Pathog. 2014 Nov 13;10(10):e1004436. doi: 10.1371/journal.ppat.1004436. eCollection 2014 Oct. No abstract available. PMID 25393405
- [Background] Capone KA, Dowd SE, Stamatas GN, Nikolovski J. Diversity of the human skin microbiome early in life. J Invest Dermatol. 2011 Oct;131(10):2026-32. doi: 10.1038/jid.2011.168. Epub 2011 Jun 23. PMID 21697884
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Costello EK, Carlisle EM, Bik EM, Morowitz MJ, Relman DA. Microbiome assembly across multiple body sites in low-birthweight infants. mBio. 2013 Oct 29;4(6):e00782-13. doi: 10.1128/mBio.00782-13. PMID 24169577
- [Background] Younge NE, Araujo-Perez F, Brandon D, Seed PC. Early-life skin microbiota in hospitalized preterm and full-term infants. Microbiome. 2018 May 31;6(1):98. doi: 10.1186/s40168-018-0486-4. PMID 29855335
- [Background] Zhu T, Liu X, Kong FQ, Duan YY, Yee AL, Kim M, Galzote C, Gilbert JA, Quan ZX. Age and Mothers: Potent Influences of Children's Skin Microbiota. J Invest Dermatol. 2019 Dec;139(12):2497-2505.e6. doi: 10.1016/j.jid.2019.05.018. Epub 2019 Aug 13. PMID 31420081
- [Background] Lehtimaki J, Karkman A, Laatikainen T, Paalanen L, von Hertzen L, Haahtela T, Hanski I, Ruokolainen L. Patterns in the skin microbiota differ in children and teenagers between rural and urban environments. Sci Rep. 2017 Mar 31;7:45651. doi: 10.1038/srep45651. PMID 28361981
- [Background] Manus MB, Kuthyar S, Perroni-Maranon AG, Nunez-de la Mora A, Amato KR. Infant Skin Bacterial Communities Vary by Skin Site and Infant Age across Populations in Mexico and the United States. mSystems. 2020 Nov 3;5(6):e00834-20. doi: 10.1128/mSystems.00834-20. PMID 33144313
- [Derived] Wilborn D, Kottner J, Hillmann K, Xu S, Konietschke F, Blume-Peytavi U. Interrelationships between Skin Structure, Function, and Microbiome of Pregnant Females and Their Newborns: Study Protocol for a Prospective Cohort Study. Dermatol Res Pract. 2021 Nov 17;2021:4163705. doi: 10.1155/2021/4163705. eCollection 2021. PMID 34840564